CLINICAL TRIAL: NCT05512780
Title: An Exploratory Clinical Study of CDK4/6 Inhibitor Dalpiciclib Combined With Letrozole in Neoadjuvant Treatment of Stage Ⅱ-Ⅲ HR-positive/HER2-negative Breast Cancer
Brief Title: Dalpiciclib Combined With Letrozole in Neoadjuvant Treatment of Stage Ⅱ-Ⅲ HR-positive/HER2-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022037
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Solid Tumor
MeSH Terms: interventions — dalpiciclib; Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dalpiciclib+ letrozole (Experimental): Dalpiciclib combined with Letrozole,28 days as one cycle.
  1. Dalpiciclib: 150 mg (p.o.) was given once daily for 3 weeks, followed by 1 week off in each 4-week cycle.
  2. Letrozole: 2.5mg, p.o., once a day, continuous administration.
  Interventions: Drug: Dalpiciclib

INTERVENTIONS:
Drug: Dalpiciclib — An exploratory study of a single-arm, open design
  All subjects enrolled will receive the following treatment:
  Dalpiciclib combined with Letrozole, 28 days as one cycle.
  Other Names: Letrozole

SUMMARY:
This is a single-arm, open-label, exploratory clinical study

DETAILED DESCRIPTION:
This is a single-arm, open-label, exploratory clinical study initiated by the investigator to evaluate the objective response rate (ORR), efficacy, and safety of Dalpiciclib combined with letrozole in the neoadjuvant treatment of stage Ⅱ-Ⅲ HR+/HER2- breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Postmenopausal women aged ≥18 years, the definition of postmenopausal:

  1. the patients with the history of bilateral oophorectomy, or age ≥ 60 years; or
  2. Age <60, natural postmenopausal state (defined as the spontaneous cessation of regular menstruation for at least 12 consecutive months, without other pathological or physiological causes), E2 and FSH at the postmenopausal levels 2. All patients were estrogen receptor (ER) positive (>10%), HER2 -negative invasive breast cancer regardless of PR expression level. Immunohistochemistry (IHC) score of 0+, or 2+ confirmed by pathology laboratory and negative in situ hybridization (ISH) test (HER-2/CEP17 ratio <2.0); 3. Treatment-naive patients with stage Ⅱ-Ⅲ tumors whose tumor staging meets the criteria of the 8th edition of the American Joint Committee on Cancer (AJCC) Staging;

Exclusion Criteria:

* 1. Received any form of anti-tumor therapy (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.) 2. Concurrently receiving any other anti-tumor therapy that those specified in the protocol; 3. Bilateral breast cancer, inflammatory breast cancer, or occult breast cancer; 4. Stage Ⅳ breast cancer;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-10 (Estimated); Primary Completion 2023-08-10 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 month
  Objective response rate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Liu Y, Yang C, Ma J, Li Y, Luo R, Han J, Wang X, Zhang Z, Ma L, Cai H, Kong X, Wang Z, Zhou X, Shi J, Zhang Y, Wang M, Wang J, Geng C. Clinical efficacy and therapy response prediction of neoadjuvant dalpiciclib plus letrozole in postmenopausal patients with HR+/HER2- stage II-III breast cancer (DARLING 01): a single-arm, open-label, exploratory study. Breast Cancer Res. 2025 Feb 13;27(1):21. doi: 10.1186/s13058-025-01976-0. PMID 39948624